CLINICAL TRIAL: NCT00605371
Title: A Pivotal, Single-Dose, Randomised, Parallel-Group, Open-Label Study to Demonstrate Bioequivalence of 250mg Lamotrigine XR Relative to 200mg + 50mg Lamotrigine XR and to Demonstrate Lack of Food Effect on 250mg Lamotrigine XR in Healthy Male and Female Volunteers
Brief Title: Bioequivalence and Food Effect of 250mg of Lamotrigine XR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEP111102
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy
Keywords: Healthy volunteers; Bioequivalence; Food Effects
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects receiving regimen A (Experimental): Eligible subjects will receive regimen A containing lamotrigine extended release tablet of 200 milligrams plus 50 milligrams in fasted state
  Interventions: Drug: Lamotrigine tablet
- Subjects receiving regimen B (Experimental): Eligible subjects will receive regimen B containing lamotrigine extended release caplet of 250 milligrams in fasted state.
  Interventions: Drug: Lamotrigine caplet
- Subjects receiving regimen C (Experimental): Eligible subjects will receive regimen C containing lamotrigine extended release caplet of 250 milligrams in fed state.
  Interventions: Drug: Lamotrigine caplet

INTERVENTIONS:
Drug: Lamotrigine tablet — Lamotrigine extended release single dose tablet will be available with dosing strengths of 200 milligrams and 50 milligrams intended to be administered orally in fasted state. It will be a round standard convex shape tablet.
  Arms: Subjects receiving regimen A
Drug: Lamotrigine caplet — Lamotrigine extended release single dose caplet will be available with dosing strength of 200 milligrams and 50 milligrams intended to be administered orally in fasted and fed state.
  Arms: Subjects receiving regimen B; Subjects receiving regimen C

SUMMARY:
This study intends to demonstrate bioequivalence and lack of food effect on 250mg lamotrigine XR in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged from 19 to 55 years, inclusive.
* Body weight >50 kg (males) or >45 kg (females) and BMI within the range 19 - 32 kg/m2 inclusive.
* Healthy as determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, vital signs and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures
* Female subjects of non-child bearing potential will be eligible to participate if they meet the following criteria:

  * Post-menopausal females defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However if indicated this should be confirmed by oestradiol and FSH levels consistent with menopause (according to local laboratory ranges).
  * Pre-menopausal females with a documented (medical report verification) hysterectomy and/or bilateral oophorectomy, the latter only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Female subjects of child bearing potential will be eligible to participate if they comply with the contraception requirements.
* A negative pre-study Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, and HIV antibody result at screening.
* A negative pre-study urine drug screen.
* A negative screen for alcohol (urine, blood or breath test).
* Signed and dated written informed consent prior to admission to the study.

Exclusion Criteria:

* Female subjects of childbearing potential will not be eligible to participate who are unwilling or unable to use an appropriate method of contraception as outlined in the inclusion criteria from at least the commencement of their last normal period prior to the first dose of study medication; and to continue until the first normal period (defined as normal for the woman, both in terms of duration and quantity of menses) after treatment or 5 half lives of the study medication, whichever is the longest .
* Female subject is pregnant (positive serum human chorionic gonadotrophin (hCG) test at screening) or lactating.
* Female subjects using hormonal contraceptive precautions including progesterone-coated IUD.
* Female subjects using oestrogen-containing hormone replacement therapy.
* Subjects who have received lamotrigine previously (subjects who received placebo in a previous study will be allowed)
* History or evidence of drug or alcohol abuse within 12 months of study start.
* QTc >450msec for women and QTc >430 msec for men on the screening 12-lead ECG.
* Current smokers of 10 or more cigarettes per day.
* History of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men within 6 months of screening. One drink is equivalent to 12 g alcohol = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Has received prescribed or non-prescribed medication (including vitamins and herbal remedies) within 14 days prior to the dosing day, which in the opinion of the Principal/Co-Investigator, may interfere with the study procedures or compromise safety.
* History of gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of clinically relevant skin rashes that, in the opinion of the investigator, might interfere with the conduct of the study.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* History of allergic, anaphylactic, hypersensitivity or idiosyncratic reaction(s) to lamotrigine or drugs of a similar type.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2008-03-06 (Actual); Study Completion 2008-03-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics ie Serum lamotrigine Cmax and AUC(0-inf) | Pre-dose and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26, 36, 48, 72, 96, 120 and 144 hours Post-dose

SECONDARY OUTCOMES:
PK (AUC (0-t), tmax and t1/2 ) | Pre-dose and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26, 36, 48, 72, 96, 120 and 144 hours Post-dose
Adverse events, changes in biochemistry, haematology, urinalysis parameters, electrocardiogram parameters, blood pressure and heart rate | Up to day 21
Serum lamotrigine AUC (0-t), tmax and t1/2 | Pre-dose and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 22, 24, 26, 36, 48, 72, 96, 120 and 144 hours Post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study LEP111102 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/LEP111102?search=study&study_ids=LEP111102#rs
- Available data/document: Informed Consent Form: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LEP111102 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register